CLINICAL TRIAL: NCT00808457
Title: Role of Chest Ultrasound in Diagnosing and Follow-up of Pneumonia. Prospective Comparison Between X-ray Chest Film in Two Planes and "Low-dose" Spiral Computed Tomography
Brief Title: Role of Chest Ultrasound in Diagnosing and Follow-up of Pneumonia
Status: Completed | Type: Observational
Sponsor: University of Jena (Other)
Responsible Party: PD Dr. med. Angelika Reißig, Pneumology, Friedrich-Schiller University Jena
Other Study IDs: 2055-06/07; PD Dr. med. Angelika Reißig; Phone: 00493641/ 9-32 41 28
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Pneumonia
Keywords: chest ultrasound; pneumonia; X-ray; CT; Sensitivity and specificity of chest ultrasound in diagnosing pneumonia
MeSH Terms: conditions — Pneumonia; Hypersensitivity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with suspected pneumonia

SUMMARY:
The study of a large number of patients (at least 200 patients) from several European centres aims to investigate the value of chest ultrasound in diagnosing and checking the course of pneumonia as compared to a chest X-ray film in two planes and - in case of a controversial X-ray finding- as compared to low-dose CT.

An X-ray finding is regarded controversial, if infiltrates cannot be reliably excluded or not reliably represented and if a definite diagnosis is, thus, not possible. A low-dose CT is indicated even in case of a positive chest ultrasound and negative X-ray finding. Sonographic recording and characterization of pneumonic infiltrates is performed both at the time of diagnosing and in the further course under therapy.

DETAILED DESCRIPTION:
The primary target criterion is

• Assessing the sensitivity of chest ultrasound in diagnosing pneumonia.

Secondary target criteria comprise

* Assessing specificity, negative and positive predictive value of chest ultrasound at the time of diagnosing,
* Characterizing pneumonic infiltrates at the time of diagnosing and further course,
* Describing the association between clinical, X-ray and sonographic findings in the course of pneumonia.

The tertiary target criterion includes

• Characterizing the range of pathogens detected by microbiological examination.

ELIGIBILITY:
Inclusion Criteria:

Patients with clinically suspected CAP who received no antibiotic treatment yet

* Patients in whom a chest X-ray in 2 planes was already performed, can be included in the study, if chest ultrasound is performed within 24 hours after X-ray and if the X-ray finding is neither available to nor known to the examiner doing the ultrasound examination.
* Age > 18 years
* Patient's declaration of consent is available.

Exclusion Criteria:

* Patients with HAP
* Age <18 years
* Patients in whom the time difference between chest ultrasound and chest X-ray in 2 planes is more than 24 hours
* Patients whose X-ray findings are with the examiner doing the ultrasound or are known to him
* Pregnancy and lactation
* Missing declaration of consent by the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically suspected community-acquired pneumonia.
Sampling Method: Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2007-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
sensitivity of chest ultrasound in diagnosing pneumonia | baseline diagnostic

SECONDARY OUTCOMES:
Specificity | baseline diagnostic

CONTACTS AND LOCATIONS:
Locations (1):
- Pneumology, Friedrich-Schiller University Jena, Jena, Thuringia, Germany

REFERENCES:
- [Background] Reissig A, Kroegel C. Sonographic diagnosis and follow-up of pneumonia: a prospective study. Respiration. 2007;74(5):537-47. doi: 10.1159/000100427. Epub 2007 Feb 27. PMID 17337882
- [Background] Copetti R, Cattarossi L. Ultrasound diagnosis of pneumonia in children. Radiol Med. 2008 Mar;113(2):190-8. doi: 10.1007/s11547-008-0247-8. Epub 2008 Apr 2. English, Italian. PMID 18386121
- [Derived] Reissig A, Mempel C, Schumacher U, Copetti R, Gross F, Aliberti S. Microbiological diagnosis and antibiotic therapy in patients with community-acquired pneumonia and acute COPD exacerbation in daily clinical practice: comparison to current guidelines. Lung. 2013 Jun;191(3):239-46. doi: 10.1007/s00408-013-9460-x. Epub 2013 Apr 6. PMID 23564195
- [Derived] Reissig A, Copetti R, Mathis G, Mempel C, Schuler A, Zechner P, Aliberti S, Neumann R, Kroegel C, Hoyer H. Lung ultrasound in the diagnosis and follow-up of community-acquired pneumonia: a prospective, multicenter, diagnostic accuracy study. Chest. 2012 Oct;142(4):965-972. doi: 10.1378/chest.12-0364. PMID 22700780